CLINICAL TRIAL: NCT04943224
Title: Optimization of the Time and Dosage of Trametinib in BRAF Negative Juvenile Patients With Refractory Histiocytosis or After the Failure of Vemurafenib Treatment
Brief Title: Optimization of the Time and Dosage of Trametinib in BRAF Negative Juvenile Patients
Acronym: TRAM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anna Raciborska (Other)
Collaborators: Maria Sklodowska-Curie National Research Institute of Oncology (Other); Łukasiewicz Research Network (Unknown); Wrocław University of Environmental and Life Sciences (Unknown)
Responsible Party: Sponsor-Investigator, Anna Raciborska, Prof Ass, Institute of Mother and Child, Warsaw, Poland
Organization: Institute of Mother and Child, Warsaw, Poland (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRAM
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Histiocytosis
Keywords: Langerhans cell histiocytosis (LCH); histiocytosis; trametinib; paediatric patients
MeSH Terms: conditions — Histiocytosis; Histiocytosis, Langerhans-Cell | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R1 time of trametinib treatment (Experimental): Patients with negative status of any mutation in ctDNA or 0-1 Disease Activity Score (DAS) in three consecutive tests in three month intervals.
  Interventions: Drug: Trametinib
- R2 time of trametinib treatment (Experimental): Patients with negative status of any mutation in ctDNA or 0-1 Disease Activity Score (DAS) in in five consecutive tests in three month intervals.
  Interventions: Drug: Trametinib

INTERVENTIONS:
Drug: Trametinib — < 6 lat 0,032mg/kg, ≥ 6 lat 0,025mg/kg,
  Other Names: Mekinist

SUMMARY:
Prospective, interventional, open, randomized, single-center, non-commercial clinical trial to optimize treatment and dosage of trametinib in juvenile patients with histiocytosis resistant to conventional therapy and without the BRAF gene mutation or after the failure of vemurafenib treatment.

DETAILED DESCRIPTION:
TRAM clinical study is part of the POLHISTIO project. The POLHISTIO project is a non-commercial clinical trial aimed at optimizing the diagnosis and treatment of juvenile patients with histiocytosis. The project objectives are defined as follows: 1) to estimate the nature and frequency of mutations in patients with histiocytosis in both tumor tissues and free-circulating DNA; 2) to compare molecular test results with clinical data; 3) to evaluate the diagnostic usefulness of the status of molecular analysis (MRD) as a prognostic factor compared with other recognized factors; 4) in the case of failure of conventional therapy - to modify treatment and to apply targeted treatment, based on molecular status of gene mutation. The project is intended to include patients from all over Poland.

ELIGIBILITY:
Inclusion Criteria:

1. Lack of mutations in the BRAF gene in tumor tissues and/or circulating tumor DNA (ctDNA) at any stage of treatment or follow-up, or failure of Vemurafenib treatment in BRAF positive patients.
2. Failure of the treatment (at least one of below needs to apply in order for this requirement to be satisfied):

   1. Progression on the I and/or II line treatment, including at least one risk organ; prior treatment should include a minimum of 6 weeks of weekly Vinblastine with a minimum of 28 days prednisolone or minimum 2 cycles of Cytosine Arabinoside in 4-day cycles and/or Cladribine in 5-day cycles as a 2nd line treatment, minimum 2 cycles, or other second-line treatment or
   2. Disease reactivation after an initial response to treatment with Vimblastine and prednisolone as the first line and/or no response to second line treatment using one of two drugs: Cytosine Arabinoside in 4- day cycles and/or Cladribine in 5-day cycles, minimum 2 cycles, or other I/ II line treatment or occurrence of involvement of at least one risk organ or

   d. Progression during Vemurafenib therapy, or e. Reactivation of disease after Vemurafenib therapy has been completed, or f. The appearance of signs of neurodegenerative disorder (ND) in MRI of the central nervous system (CNS).
3. Signing of informed consent for trial participation (including for Trametinib treatment) according with current legal regulations.
4. Consent to the use of effective contraception throughout the Trametinib administration period and a minimum of 1 year after discontinuation in patients at puberty and sexual maturity.
5. Participation in HISTIOGEN trial.

Exclusion Criteria:

1. Lack of inclusion criteria.
2. Pregnancy and breastfeeding .
3. Hypersensitivity to the study drug or any of its ingredients.
4. Iritis, uveitis, obstruction of the retinal veins.
5. Simultaneous treatment with other drugs which might interact with Trametinib.
6. Persistent toxicity related to prior therapy, making it impossible to treat with Trametinib.
7. Diagnosis of other malignancies before study inclusion.
8. Other acute or persistent disorders, behaviors or abnormal laboratory test results, which might increase the risk related to the participation in this clinical trial or to taking the study drug, or which might influence the interpretation of the study results, or which, in the investigator's opinion, disqualify a patient from participating in the trial.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 2 years
  Event-free survival (EFS) was defined as the time interval from the date of diagnosis to the date of disease progression, recurrence, second malignancy, death or to date of last follow-up for patients without events.

SECONDARY OUTCOMES:
Molecular relapse (in ct DNA) | 2 years
  Molecular relapse was defined as the time interval from the date of any mutation negativization to the date of positive results of any mutation
Time to negative mutation test results (in ct DNA) | 2 years
  Time to negative mutation test results (in ct DNA) was defined as the time interval from the date of positive mutation to the date of negative results of any mutation

CONTACTS AND LOCATIONS:
Overall Officials: Anna Raciborska, Principal Investigator — Mother and Child Institute
Locations (1):
- Mother and Child Institute, Warsaw, Mazovian, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardoso E, Mercier T, Wagner AD, Homicsko K, Michielin O, Ellefsen-Lavoie K, Cagnon L, Diezi M, Buclin T, Widmer N, Csajka C, Decosterd L. Quantification of the next-generation oral anti-tumor drugs dabrafenib, trametinib, vemurafenib, cobimetinib, pazopanib, regorafenib and two metabolites in human plasma by liquid chromatography-tandem mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2018 Apr 15;1083:124-136. doi: 10.1016/j.jchromb.2018.02.008. Epub 2018 Feb 8. PMID 29544202
- [Background] Cox DS, Allred A, Zhou Y, Infante JR, Gordon MS, Bendell J, Jones S, Burris H 3rd, Orford K. Relative bioavailability of pediatric oral solution and tablet formulations of trametinib in adult patients with solid tumors. Clin Pharmacol Drug Dev. 2015 Jul;4(4):287-94. doi: 10.1002/cpdd.152. Epub 2014 Oct 27. PMID 27136909
- [Background] Crombag MBS, van Doremalen JGC, Janssen JM, Rosing H, Schellens JHM, Beijnen JH, Steeghs N, Huitema ADR. Therapeutic drug monitoring of small molecule kinase inhibitors in oncology in a real-world cohort study: does age matter? Br J Clin Pharmacol. 2018 Dec;84(12):2770-2778. doi: 10.1111/bcp.13725. Epub 2018 Sep 26. PMID 30068020
- [Background] Farnault L, Helias-Rodzewicz Z, Venton G, Fanciullino R, Gabriel S, Mescam L, Haroche J, Donadieu J, Emile JF. Response to trametinib of histiocytosis with an activating PTPN11 mutation. Leuk Lymphoma. 2020 Jan;61(1):194-197. doi: 10.1080/10428194.2019.1650175. Epub 2019 Aug 8. No abstract available. PMID 31393194
- [Background] Herbrink M, de Vries N, Rosing H, Huitema ADR, Nuijen B, Schellens JHM, Beijnen JH. Development and validation of a liquid chromatography-tandem mass spectrometry analytical method for the therapeutic drug monitoring of eight novel anticancer drugs. Biomed Chromatogr. 2018 Apr;32(4). doi: 10.1002/bmc.4147. Epub 2017 Dec 19. PMID 29165815
- [Background] Infante JR, Fecher LA, Falchook GS, Nallapareddy S, Gordon MS, Becerra C, DeMarini DJ, Cox DS, Xu Y, Morris SR, Peddareddigari VG, Le NT, Hart L, Bendell JC, Eckhardt G, Kurzrock R, Flaherty K, Burris HA 3rd, Messersmith WA. Safety, pharmacokinetic, pharmacodynamic, and efficacy data for the oral MEK inhibitor trametinib: a phase 1 dose-escalation trial. Lancet Oncol. 2012 Aug;13(8):773-81. doi: 10.1016/S1470-2045(12)70270-X. Epub 2012 Jul 16. PMID 22805291
- [Background] Lian T, Li C, Wang H. Trametinib in the treatment of multiple malignancies harboring MEK1 mutations. Cancer Treat Rev. 2019 Dec;81:101907. doi: 10.1016/j.ctrv.2019.101907. Epub 2019 Oct 14. PMID 31715422
- [Background] Lorillon G, Jouenne F, Baroudjian B, de Margerie-Mellon C, Vercellino L, Meignin V, Lebbe C, Vassallo R, Mourah S, Tazi A. Response to Trametinib of a Pulmonary Langerhans Cell Histiocytosis Harboring a MAP2K1 Deletion. Am J Respir Crit Care Med. 2018 Sep 1;198(5):675-678. doi: 10.1164/rccm.201802-0275LE. No abstract available. PMID 29694792
- [Background] Nelson DS, van Halteren A, Quispel WT, van den Bos C, Bovee JV, Patel B, Badalian-Very G, van Hummelen P, Ducar M, Lin L, MacConaill LE, Egeler RM, Rollins BJ. MAP2K1 and MAP3K1 mutations in Langerhans cell histiocytosis. Genes Chromosomes Cancer. 2015 Jun;54(6):361-8. doi: 10.1002/gcc.22247. Epub 2015 Mar 31. PMID 25899310
- [Background] Ouellet D, Kassir N, Chiu J, Mouksassi MS, Leonowens C, Cox D, DeMarini DJ, Gardner O, Crist W, Patel K. Population pharmacokinetics and exposure-response of trametinib, a MEK inhibitor, in patients with BRAF V600 mutation-positive melanoma. Cancer Chemother Pharmacol. 2016 Apr;77(4):807-17. doi: 10.1007/s00280-016-2993-y. Epub 2016 Mar 3. PMID 26940938